CLINICAL TRIAL: NCT05604833
Title: The Effect of Progressive Muscle Relaxation Exercises on Sleep Quality in Patients Receiving Hemodialysis Treatment: A Randomized Controlled Study
Brief Title: Measuring Sleep Quality With Puki in Hemodialysis Patients Performing Progressive Muscle Relaxant Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KARATAY.halime.hakverir1
Record Dates: First submitted 2022-10-16; First posted 2022-11-03 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: A Randomized Controlled Study
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding Due to the characteristics of the study, blinding cannot be applied to the participants. In order to eliminate the bias, the data of the study will be collected and recorded by an impartial researcher (assistant researcher) who does not know the groups trained by the researcher. The statistics of the research will be carried out by an independent statistician who does not know the groups. In this way, the prevention of bias will be ensured.
  The implementation phase of the research is indicated in Table 1 The Implementation Phases of the Research and the Consort diagram (Figure 1. Consort Scheme).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): they will November progressive muscle relaxation exercise
  Interventions: Behavioral: Progressive Muscle Relaxation Exercises
- no ıntervention (No Intervention): to be followed without exercise

INTERVENTIONS:
Behavioral: Progressive Muscle Relaxation Exercises — In the research, data will be collected with the "Descriptive Information Form" and "Pittsburgh Sleep Quality Index (PUKI)". Statistical analysis of the data obtained as a result of the research will be made in the IBM SPSS25 program. This study was planned because it is thought that making progressive muscle relaxation exercises (PKGE) in patients with poor sleep quality who receive hemodialysis treatment will be effective in increasing sleep quality, since it is easy to learn, can be done anywhere, and has no side effects.
  Arms: experimental

SUMMARY:
Chronic kidney disease is a chronic disease that negatively affects the quality of life of individuals, physically, socially and psychologically. Although the problems due to kidney failure are brought under control with hemodialysis treatment, the continuation of the treatment depending on the machine and the difficulties brought by the treatment process cause the patient to experience many negativities, especially insomnia and fatigue. Studies have shown that the prevalence of insomnia in patients receiving hemodialysis treatment is high and sleep problems are seen in 40-83% of them, the quality of sleep is low, and the quality of life is adversely affected by this situation, and the mortality rate increases. This study will be conducted to evaluate the effect of progressive muscle relaxation exercises on sleep quality applied to individuals receiving hemodialysis treatment for chronic kidney disease (CKD) and having poor sleep quality. The research will be conducted as a randomized controlled trial with patients receiving hemodialysis treatment at Private Nephrotrans Karatay Dialysis Center between March and September 2022. The sample size of the study was determined according to the results of a similar study using the G*Power 3.1., 9.7 program with α = 0.05 and 90% power. The sample number was determined as 80 patients, including experimental (n=40) and control (n=40). In the research, data will be collected with the "Descriptive Information Form" and "Pittsburgh Sleep Quality Index (PUKI)". Statistical analysis of the data obtained as a result of the research will be made in the IBM SPSS25 program. This study was planned because it is thought that making progressive muscle relaxation exercises (PKGE) in patients with poor sleep quality who receive hemodialysis treatment will be effective in increasing sleep quality, since it is easy to learn, can be done anywhere, and has no side effects.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a chronic disease that negatively affects the quality of life of people in physical, social and psychological terms, although it is an important public health problem that is common in the world and in our country. Chronic kidney disease is defined as a chronic and progressive deterioration in the fluid-solute balance and metabolic-endocrine functions of the kidney with a permanent decrease in the glomerular filtration rate . Patients with a GFR below 5-10 ml/min need renal replacement therapy. Renal replacement therapy is defined as a form of treatment that performs kidney function due to the inability of the kidneys to perform their normal blood filtering function. The number of patients in need of renal replacement therapy in our country is increasing day by day. In the early stages of CKD, RRT is needed due to the inability to control the disease with diet and drug therapy. Renal replacement therapies are performed in the form of hemodialysis, peritoneal dialysis and transplantation. Hemodialysis is the most preferred renal replacement therapy method in the treatment of CKD in our country. It is aimed to reduce mortality and morbidity rates by increasing the quality of life of patients with hemodialysis treatment. Hemodialysis is the process of cleaning the blood and returning it to the patient by passing the blood taken from the appropriate vascular access path to the patient through a dialyzer (filter) with a semi- permeable structure with the help of a dialysis machine to remove substances that cannot be excreted from the body, such as urea, creatinine, phosphorus, due to the inability of the kidney to perform its functions. Although the problems that develop due to kidney failure are controlled by hemodialysis treatment, the treatment is continued depending on the machine and the difficulties caused by the treatment process cause the sick person to experience many negativities, especially insomnia, fatigue. The etiology of insomnia observed in dialysis patients is based on many factors. Biochemical and metabolic changes, lifestyle, depression, anxiety, and other underlying sleep disorders all have an impact on the development of chronic sleep disorders. Insomnia is characterized by symptoms that indicate poor sleep quality, such as inability to fall asleep on time, involuntary waking up at night, failure to get up rested in the morning, disruption of daytime functions along with daytime napping. Studies have shown that the prevalence of insomnia is high in patients receiving hemodialysis treatment, and 40-83% have sleep problems, poor sleep quality, and this negatively affects the quality of life, cognitive impairment, inattention increases, work efficiency decreases, and causes an increase. In a study conducted by Yıldırım and his colleagues on insomnia, they found that almost all of the patients undergoing hemodialysis had sleep problems the night before dialysis (95.5%) and the night after (93.6%). In studies, there are studies that show that relaxation exercises are useful for eliminating sleep problems and improving sleep quality in patients receiving hemodialysis treatment. In a study conducted by Amini and colleagues, it was found that progressive muscle relaxation exercises applied before going to bed at night for 60 days improved sleep quality. Also in a study of Maryam and his other friends, who are on hemodialysis treatment to patients in days once, and once at night before going to bed twice a day progressive relaxation progressive relaxation exercise for 30 days in a survey commissioned by Nov Nov exercises a positive impact on sleep quality in patients who are on hemodialysis (HD) treatment was shown to provide. Relaxation is a method that reduces arousal before going to sleep. When relaxation exercises are performed regularly in accordance with the rule by providing an appropriate environment, tension, stress effects, blood pressure and heart rate decrease, attention is diverted to patients; sleep pain, etc. it is stated in the studies that it is effective in solving the problem. Relaxation techniques are practices that reduce stress symptoms, provide physical awareness, increase focus, calm down, and reduce physiological hypersensitivity due to sleep disturbance. In addition, relaxation exercises contribute to improving the quality of life of the individual and maintaining his general health. Relaxation exercises deep breathing exercises, meditation, progressive November muscle relaxation exercises are exercises such as progressive November muscle relaxation exercises, was founded in 1929 by Dr. It was developed by Jacopson. Nov progressive relaxation exercises, Nov individually by the contraction and relaxation groups, a simple process without the feeling of pain and tension is defined as. Progressive November relaxation exercises November relaxation exercises can also be defined as a type of exercise that allows people to relax in moments of tension, by contracting and relaxing muscle groups from the face to the feet. Nov progressive relaxation exercises are easy to learn, can be done anywhere and side effects during treatment of hemodialysis patients whose sleep quality is poor in the absence of progressive relaxation exercises are thought to be effective in improving quality of sleep be made of Nov.

1.1. Purpose Of The Study This study was planned to evaluate the effect of progressive muscle relaxation exercises (PC November) on sleep quality in patients receiving hemodialysis treatment. 2. GENERAL INFORMATION 2.1. Hemodialysis Hemodialysis treatment of end-stage kidney disease in patients with creatinine, urea from the blood of substances that cannot be removed from the patient and breathe with the help of machine fluid of the blood of the contents of a semi-permeable membrane by virtue of the dialysis fluid is passed into and reorganization of given back to the patient. According to the 2020 records of the Turkish Society of nephrology, 11,596 patients started renal replacement therapy in our country in 2020, of which 9,081 were patients receiving hemodialysis treatment, accounting for 76%. Hemodialysis is the most preferred renal replacement therapy in the treatment of chronic kidney disease. With this form of treatment, it is aimed to increase the quality of life and survival of patients, as well as to reduce mortality and morbidity rates. High compliance with treatment prolongs the life expectancy of patients. Patients who are on hemodialysis (HD) treatment for fatigue, Nov cramps, depression, nausea, vomiting, hypotension, sleep problems, irritability, itching, bone pain,and dryness of the skin, constipation, diarrhea, sexual inability, physical and psychological symptoms such as mood disorders are observed. Patients experience difficulties in daily living activities and social life related to the symptoms they experience. Pharmacological and nonpharmacological methods are used to cope with these symptoms faced by patients. Although patients undergo regular dialysis, they experience difficulty in complying with high fluid intake, medication and diet between two dialysis sessions Dec. It is easier for patients to cope with the disease and symptoms with the educational support, effective nursing care, individual support provided. 2.2. Quality of Sleep Covering a third of our lives, sleep is essential for physical, emotional and cognitive health. Sleep is defined as a period of renewal that allows the organism to rest, during which the immune system continues to work, frees the individual from complex thoughts with a state of unconsciousness that has a return, and re-prepares the body for life. Sleep, which is one of the basic human needs, is important at every stage of the development period. It is defined as the quality of sleep that an individual feels fit, rested after waking up, that his night sleep is not interrupted, that he feels energetic to live the new day.

The quality of sleep is physical (age, gender, physical activity, medication use, emotional status, etc.) and environmental (the fact that the environment is bright, heat, sound, etc.) factors influence. Conditions such as decreased attention, fatigue, depression, irritability, drowsiness, cognitive disorders, increased sensitivity to pain, as well as deterioration in motivation, emotion and thinking of individuals with poor sleep quality are observed.

Studies conducted in hemodialysis patients indicate a high prevalence of sleep problems. Sleep problems are counted as napping during the day, difficulty falling asleep at night, frequent awakenings. In addition, it can lead to sleep problems for reasons such as anxiety, itching, depression related to the disease. For this reason, in nursing applications (evaluating sleep habits, preventing him from sleeping during the day, exercise, aramotherapy, etc.) care should be provided with the aim of identifying sleep problems early and improving sleep quality. 2.3. Progressive November Muscle Relaxation Exercises Relaxation means relaxation, rest. Progressive muscle relaxation exercises were first introduced in November 1929 by Dr. It is a form of treatment developed and described by Edmund Jacobson as cognitive behavioral techniques that allow muscles to November and relax voluntarily. Regular performance of relaxation exercises activates the parasympathetic system and provides hemoostatic balance. PK November, with a calm mind, muscles relax, tension disappears and anxiety decreases. Progressive relaxation exercises have benefits such as reducing the individual's sensitivity to stress, tension, fatigue, facilitating the transition to sleep, improving the quality of life. The main purpose of relaxation exercises is that individuals can achieve relaxation on their own in moments of tension by understanding the difference in muscle tension November and relaxation. During November, the muscles in the hands, arms, neck, shoulders, face, chest, hips, thighs, feet and fingers contract and relax. Voice recordings lasting an average of 30 minutes are listened to and exercise is performed in a comfortable and calm environment.

In the meta-analysis conducted by Yang et al., it was found that patients who perform progressive muscle relaxation exercises improve the quality of sleep, relieve negative emotions, improve the quality of life by November by improving psychological functions. Progressive muscle relaxation exercises, which are a non pharmacological intervention method, have been widely used to relieve anxiety November and pain. According to meta-analysis, pror November relaxation exercises provided positive relief from fatigue, sleep problems and mood in hemodialysis patients. 3. MATERIALS AND METHODS In this section, information will be given about the form of the research, the time and place of the research. 3.1. The Form of the Research

A randomized controlled trial was planned to evaluate the effect of progressive muscle relaxation exercises (PC November) on sleep quality in patients receiving hemodialysis treatment. 3.2. Place and Time of Research November February 10, 2022- February 20, 2023 the research will be conducted at the private Nephrotrans Karatay Dialysis Center. In the center hemodialysis, a total of 50+1(spare) has a dialysis machine, central 2 doctors and 2 nurses, 4 emergency medical technicians (ATT), 9 dialysis technician with 3 sessions daily (morning-afternoon-evening) in the form of six days a week, serving a total of 218 patients. It is planned that there will be a health worker (nurse, ATT, dialysis technician) for 6 patients in each dialysis session. Before the patient is placed on dialysis, the amount of liquid to be drawn is weighed and calculated according to his dry weight. While the patient is on dialysis, bleeding control is carried out without fail, the patient is given information about education about bleeding and to report when a problem with bleeding develops. In addition, complications that may occur during and after hemodialysis (nausea, vomiting, hypotension, November cramps, etc.).) patient / patient relatives training is carried out on the subject. Before the patient is placed on dialysis, vital signs are taken, vascular access path control is performed, the patient whose vital signs are at normal values and there are no problems in the vascular access path is taken to dialysis treatment. What should the patient pay attention to during dialysis (do not cover and lie on the arm that has a fit, nausea, cramps occur during dialysis, hypotension, fever or chills, etc. in this case, the nurse is informed about the information). In addition, the patient is informed about the vascular access route bleeding control at the end of the dialysis session and that he may feel tired, weak at the end of dialysis, and that he should call the dialysis center when there are any problems at home. If the dialysis center meets the route, the patient has the opportunity to choose the appropriate one from the morning lunch and evening sessions. 3.3. The Universe and Sample of the Research The research universe will consist of 218 patients at the private Nephrotrans Karatay Dialysis Center, where the research will be conducted. The number of samples of the research, G*Power 3.1., determined according to the results of a similar study using the 9.7 program with α = 0.05 and 90% power. 32 to 64 in each group participant is calculated as the sample, and by considering the potential losses during operation this number to 40 participants for each group was 80. 3.3.1. Criteria for Inclusion in the Study 18 years of age or older Pittsburgh Sleep Quality Index (PUKI) score of 5 points and above, Who has been receiving hemodialysis treatment for at least 3 months, Convenient to upload progressive November muscle relaxation exercise video to the mobile phone located Who volunteered to participate in the research

3.3.2. Criteria for Non-Inclusion in the Study Hearing impaired Who has a physical disability to perform relaxation exercises Depression, schizophrenia, etc. with a diagnosis of psychiatric illness Relaxation exercise (yoga, breathing and meditation, etc.) for the last six months.) acting 3.3.3. Termination Criteria

• Who did not practice relaxation exercises for at least 2 consecutive days and 9 days a month in total during the research process, Transfer from the center where the research was conducted to another center for dialysis treatment,

3.4. Variables of the Research

ındependent Variable: Progressive muscle relaxation exercises (PK November) Dependent Variable: Sleep quality and sleep quality sub- dimensions (sleep latency (delay), habitual sleep efficiency, sleep disturbance, use of sleeping medications and daytime dysfunction)

3.5. Research Hypothesis H1: The total PKI score of patients receiving hemodialysis treatment and performing progressive muscle relaxation exercises (PKGE) is lower than the total PKI score of patients who do not perform PKGE November 3.6. Data Aggregate Tools and Data Collection The data will be collected with the "Introductory Information Form" and the "Pittsburgh Sleep Quality Index 3.6.1. Data Collection Tools In the study, the data will be collected using the Introductory Information Form, Pittsburgh Sleep Quality Index (PSQI). 3.6.1.1. Introductory Information Form It consists of a total of 14 questions in which the participants' age, gender, education, marital status, profession and illness and information developed by the researchers using the literature were evaluated. (Additional.1 Introductory Information Form) 3.6.1.2. Pittsburgh Sleep Quality Index It is a self-reported assessment tool developed by Buysse and colleagues that provides information about the quality of sleep and the type and severity of sleep disorders in the last month. The validity and reliability of PUKI, which provides an assessment of the quality, quantity, presence and severity of sleep disorders in an individual and contains 19 questions, was performed in Turkish by Ağargün. The PUKI consists of seven items in which subjective sleep quality, sleep delay, sleep duration, sleep efficiency, sleep disturbance, use of sleeping pills and deterioration in daytime work are evaluated. The response of each of them is scored between 0-3 according to the frequency of symptoms. Dec. Scoring is made as 0 if it has never happened during the last month, 1 if it is less than once a week, 2 if it is once or twice a week, 3 if it is three or more times a week. The sleep quality assessment asked in the questionnaire is scored as very good 0, very good 1, very bad 2, very bad 3. The global score obtained ranges from 0-21, and high values indicate that the quality of sleep is poor and the level of sleep disturbance is high. Dec. A global score of 5 or above clinically indicates that sleep quality is significantly poor.

3.7. Application of Research 3.7.1 Randomization : Randomizasyon.org groups from the site will be randomized by the block randomization method by a person who knows the research other than the researcher. The numbers in the randomization list will be placed in closed envelopes in order. After the consent of the patients who meet the criteria for admission to the study is obtained and the preliminary tests are completed, their appointments will be made according to this list. 3.7.2. Blinding Due to the characteristics of the study, blinding cannot be applied to the participants. In order to eliminate the bias, the data of the study will be collected and recorded by an impartial researcher (assistant researcher) who does not know the groups trained by the researcher. The statistics of the research will be carried out by an independent statistician who does not know the groups. In this way, the prevention of bias will be ensured.

The implementation phase of the research is indicated in Table 1 The Implementation Phases of the Research and the Consort diagram (Figure 1. Consort Scheme).

ELIGIBILITY:
Inclusion Criteria:

* 3.3.1. Criteria for Inclusion in the Study

  * who are 18 years of age or older, *
  * Pittsburgh Sleep Quality Index (PUKI) score of 5 points and above,
  * Who has been receiving hemodialysis treatment for at least 3 months,
  * Convenient to upload progressive November muscle relaxation exercise video to the mobile phone located
  * Who volunteered to participate in the research

Exclusion Criteria:

* 3.3.2. Criteria for Non-Inclusion in the Study

  * Hearing impaired
  * Who has a physical disability to perform relaxation exercises
  * Depression, schizophrenia, etc. with a diagnosis of psychiatric illness
  * Relaxation exercise (yoga, breathing and meditation, etc.) for the last six months.) acting

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Sleep Quality | two months
  measuring the effect of progressive November relaxation exercise on sleep quality

CONTACTS AND LOCATIONS:
Locations (1):
- KTO Karatay Üniversitesi, Konya, Turkey (Türkiye)